CLINICAL TRIAL: NCT06345989
Title: Time and Cost-implications of Intraoral Scans Vs Alginate Impressions: a Randomised Controlled Trial
Brief Title: Time and Cost-implications of Intraoral Scans Vs Alginate Impressions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 187157; 340246 (Registry Identifier: Integrated Research Application System)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-12

CONDITIONS: Alginate Impression; Intraoral Scanner; Time; Cost
Keywords: Orthodontics; Alginate; Impression; Intraoral; Scanner

STUDY DESIGN:
Intervention Model Description: Prospective single-centre parallel arm randomised controlled trial, with an allocation ratio of 1:1 to investigate the difference in chairside time and cost of alginate impressions vs intraoral scans.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, blinding to intervention will not be possible for the participants or clinicians during data acquisition. All data analysis will be carried out blinded using a coded data set.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alginate impression (Active Comparator): Alginate impression
  Interventions: Procedure: Alginate impression
- Intraoral scan (Active Comparator): Intraoral scan using Trios 3Shape Scanner
  Interventions: Procedure: Intraoral scan

INTERVENTIONS:
Procedure: Alginate impression — Alginate impressions are a traditional method for creating dental moulds which are used in orthodontic records. Plastic trays are sized to fit the upper and lower jaws, and the alginate is mixed into a putty before being placed in the trays. The putty is then used to take detailed impressions of the patient's teeth. To capture an accurate bite registration, the patient bites down on a piece of warmed wax.
  Arms: Alginate impression
Procedure: Intraoral scan — Intraoral scanners capture multiple images of the mouth, which are combined to create a three-dimensional model of the patient's upper and lower teeth. The scanning wand is passed methodically over the surface of the teeth to gather all the necessary information, which is displayed in real-time on a computer screen.
  Arms: Intraoral scan

SUMMARY:
BACKGROUND: Alginate impressions have long been a staple in orthodontics, but with recent technological advancements, digital impressions via intraoral scans are gaining increasing popularity. While much research has focused on patient preference and the accuracy of these techniques, there is a notable gap in the literature regarding chair side time and associated costs. Existing studies on chair side time comparisons between alginate impressions and intraoral scanning yield inconsistent results, underscoring the need for further investigation. This study aimed to evaluate the chair side time and cost implications of intraoral scanning and alginate impressions.

OBJECTIVES: The primary objective is to compare the chair side time taken for alginate impressions and intraoral scanning of orthodontic patients aged 9 years and over in an orthodontic department at a district general hospital. The secondary objective is to evaluate the costs associated with alginate impressions and intraoral scanning of orthodontic patients described above.

DESIGN, SETTING AND PARTICIPANTS: A prospective, single-centre, parallel-arm randomised controlled trial (1:1 allocation) to be undertaken in a district general hospital. Sixty-eight orthodontic patients aged nine and above, requiring study models, will be recruited during new patient appointments at the Orthodontic Department at Queen's Medical Centre, Nottingham. Patients will be randomly assigned to either the intraoral scan or alginate impression group, with chair side time recorded for each procedure, including retakes. The IOS group will use the 3Shape TRIOS scanner, while the alginate group will follow standard procedures. The costs of each technique will be calculated following the procedure. Ethical approval was obtained from a Health Research Authority Research Ethics Committee.

OUTCOMES: N/A

CONCLUSIONS: N/A

DETAILED DESCRIPTION:
RATIONALE: This research project investigates the evolving landscape of orthodontic practices by comparing the time and cost implications of two prevalent techniques: intraoral scanning and traditional alginate impressions.

Whilst the majority of the existing literature reveals patient preference in favour of intraoral scanning, it remains common practice to use alginate impressions for orthodontic records. Considerations such as time implications, device costs, associated software expenses, and the need for clinician training pose challenges to widespread adoption of intraoral scanning. When comparing chairside time taken for intraoral scans versus alginate impressions, there are inconsistent findings, necessitating a comprehensive investigation.

The outcomes of this study will provide crucial insights into the practicality and economic viability of intraoral scanning versus alginate impressions in orthodontic settings, thereby informing clinical practices and facilitating technological assimilation within the United Kingdom. This research contributes to strengthening the evidence base surrounding orthodontic techniques and their implications for patient-centred care.

DESIGN: Prospective single-centre parallel-arm randomised controlled trial, with an allocation ratio of 1:1, to investigate the difference in chair side time and cost of alginate impressions vs intraoral scans.

SETTING: A single-centre study was undertaken in the Orthodontic Department at Queens Medical Centre (QMC), Nottingham University Hospitals NHS Trust.

EXCLUSION CRITERIA:

* Patients who will not be undergoing orthodontic treatment in secondary care (referral back to primary care).
* Patients who refuse to consent to inclusion in the trial.
* Patients with contraindications to either impression method (e.g., severe gag reflex, claustrophobia, medical history that would preclude the taking of dental impressions).
* Patients with severe dental anxiety.
* Patients with cleft lip and/or palate.

RECRUITMENT: Orthodontic patients aged 9 years and above attending the orthodontic department at Nottingham University Hospital for a new patient assessment will be assessed by an appropriately trained clinician for their eligibility for inclusion in the trial.

CONSENT: The Chief Investigator (CI) retains overall responsibility for the conduct of research, including the taking of informed consent of patients. The CI must ensure that any person delegated responsibility to participate in the informed consent process is duly authorised, trained and competent to participate according to the ethically approved protocol, principles of Good Clinical Practice (GCP) and Declaration of Helsinki.

The clinician will carry out a screening process consisting of a written checklist to assess whether patients meet the inclusion criteria. Following the identification of eligible patients, the trial will be discussed in more detail with the potential patient and/or their parent/guardian. Discussion of the trial will be undertaken by a clinician trained in the REC-approved research protocol. The discussion will involve the following:

* Introduction

  * An explanation to the patient and their parent/guardian as to the purpose and the nature of the research
  * An outline of what the research involves.
* Involvement

  o What would be required by the patient / their child.
* Benefits

  * Discussion of any potential benefits that may be involved.
* Risks o Discussion of any potential risks that may be involved.
* Alternatives

  o Discussion of the alternative options should the patient and/or their parent/guardian not want to take part in the trial.
* Withdrawal

  * Should the patient and/or their parent/guardian wish to withdraw from the study, they may do so at any time and do not have to give a reason as to why they are withdrawing.
  * It will be emphasised that should the patient and/or their parent/guardian choose to withdraw from the study, this will not impact the care they receive.
* Questions

  o The patient and/or their parent/guardian will be allowed to ask any questions they may have related to the trial.
* Capacity

  * The capacity of the patients shall be assessed.
  * Patients over the age of 16 may consent to inclusion in the trial should they have the capacity to do so.
* Contact o Information regarding a point of contact for the trial will be given to the patient and/or their parent/guardian.

Any patients who meet the exclusion criteria will not be included in the trial. Following a verbal discussion of the trial, the patient and/or their parent/guardian will be provided with a patient information sheet and given the opportunity to ask any questions before deciding if they would provisionally like to enrol in the trial.

At the beginning of the next visit, the patient's and/or their parent's/guardian's consent to inclusion in the trial will be confirmed. Should the patient and/or their parent/guardian consent to inclusion, the patient will be enrolled in the trial and randomly allocated to a treatment group (either alginate impression or intraoral scan). Informed consent must be obtained before the patient undergoes procedures that are specifically for the trial.

Should the patient and/or their parent/guardian decline to participate in the trial, they will continue with their normal orthodontic treatment and not receive any further information regarding the trial. For children under the age of 16 years, assent will be sought from their parent/guardian. Adults who are unable to consent will not be included in the trial.

Should a patient and/or their parent/guardian wish to withdraw from the trial, they may do so at any point and do not have to stipulate as to why. Patients and/or their parents/guardians will be reassured that withdrawal from the trial will not affect their treatment.

Refusal from the patient to take part in the trial must be respected, and no reason is required. Patients remain free to withdraw from the trial at any time without stipulating why and without prejudicing their further treatment. Patients must be provided with a contact point where they may obtain further information about the trial. Data collected up to the point of withdrawal can only be used after withdrawal if the patient has consented to this.

TRIAL: Once consent has been gained and the patient has been randomly allocated to a treatment group, one of the following procedures will be followed:

Intraoral scanner group

* The 3Shape TRIOS unit will be set up, tip warmed, and patient details entered into the system.
* Timer started: A timer will be started by the dental nurse when the 3Shape TRIOS unit is removed from the holder by the clinician.
* The clinician will complete the scan in the order on the system (lower arch, upper arch and bite registration) and save it to the system.
* Timer stopped: Once the scan taken is of good quality, the clinician will place the 3Shape TRIOS unit back in the holder, and the dental nurse will stop the timer.
* The clinician will check the quality of the scan against example photos, which will demonstrate good quality scans. If the scan does not meet these quality standards, it will require a retake. If any retakes are required, the timer will be resumed, and the procedure will be carried out as above.
* The time taken for the procedure and the number of retakes required will be recorded in the data collection section of the case report form (CRF).

Alginate impression group

* The clinical area will be set up with the appropriate equipment- alginate, water, mixing bowl, spatula, measuring cup, upper and lower trays, adhesive and wax.
* The clinician will check the appropriate tray sizes for the patient.
* The timer started: A timer will be started by the dental nurse when the water for the alginate impression is poured into the mixing bowl.
* The upper and lower impressions will be taken.
* A wax bite registration will then be taken.
* Timer stopped: The timer will be stopped by the dental nurse when the bite registration is removed from the patient's mouth and placed in the designated area on the worktop.
* The clinician will check the quality of the impressions and bite registration against example photos, which will demonstrate good quality impressions/bite registration. If the impressions or bite registration does not meet these quality standards, then they will require a retake. If any retakes are required, the timer will be resumed, and the procedure will be carried out as above.
* The time taken for the procedure, a number of scoops of alginate used and the number of retakes required will be recorded in the data collection section of the CRF.

Measurements taken will only include the chairside time taken to make the impression and will not include time taken for disinfection and processing of impressions.

ANALYSES: Tests for normality will be used to determine whether the data is normally distributed. If the data is normally distributed and with equal variances between the two groups, then a two-sided independent t-test will be used. If the data is not normally distributed, a Mann-Whitney U test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients aged 9 years and above requiring study models, having attended the orthodontic department at Nottingham University Hospitals for a new patient assessment.

Exclusion Criteria:

* Patients who will not be undergoing orthodontic treatment in secondary care (referral back to primary care).
* Patients who refuse to consent to inclusion in the trial.
* Patients with contraindications to either impression method (e.g., severe gag reflex, claustrophobia, medical history that would preclude the taking of dental impressions).
* Patients with severe dental anxiety.
* Patients with cleft lip and/or palate.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Chairside time taken for alginate impressions vs intraoral scans. | 12 months
  To compare the mean chairside time taken for alginate impression taking and intraoral scanning of orthodontic patients aged 9 years and over, in an orthodontic department at a district general hospital.

SECONDARY OUTCOMES:
Cost implications of alginate impressions vs intraoral scans. | 12 months
  Evaluation of the costs associated with alginate impressions and intraoral scanning of orthodontic patients described above.

CONTACTS AND LOCATIONS:
Overall Officials: Norah Flannigan, Study Chair — University of Sheffield
Locations (1):
- Queens Medical Centre, Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bosoni C, Nieri M, Franceschi D, Souki BQ, Franchi L, Giuntini V. Comparison between digital and conventional impression techniques in children on preference, time and comfort: A crossover randomized controlled trial. Orthod Craniofac Res. 2023 Nov;26(4):585-590. doi: 10.1111/ocr.12648. Epub 2023 Mar 20. PMID 36891891
- [Background] Burhardt L, Livas C, Kerdijk W, van der Meer WJ, Ren Y. Treatment comfort, time perception, and preference for conventional and digital impression techniques: A comparative study in young patients. Am J Orthod Dentofacial Orthop. 2016 Aug;150(2):261-7. doi: 10.1016/j.ajodo.2015.12.027. PMID 27476358
- [Background] Burzynski JA, Firestone AR, Beck FM, Fields HW Jr, Deguchi T. Comparison of digital intraoral scanners and alginate impressions: Time and patient satisfaction. Am J Orthod Dentofacial Orthop. 2018 Apr;153(4):534-541. doi: 10.1016/j.ajodo.2017.08.017. PMID 29602345
- [Background] Christopoulou I, Kaklamanos EG, Makrygiannakis MA, Bitsanis I, Tsolakis AI. Patient-reported experiences and preferences with intraoral scanners: a systematic review. Eur J Orthod. 2022 Jan 25;44(1):56-65. doi: 10.1093/ejo/cjab027. PMID 34089258
- [Background] Glisic O, Hoejbjerre L, Sonnesen L. A comparison of patient experience, chair-side time, accuracy of dental arch measurements and costs of acquisition of dental models. Angle Orthod. 2019 Nov;89(6):868-875. doi: 10.2319/020619-84.1. Epub 2019 Jul 1. PMID 31259615
- [Background] Grunheid T, McCarthy SD, Larson BE. Clinical use of a direct chairside oral scanner: an assessment of accuracy, time, and patient acceptance. Am J Orthod Dentofacial Orthop. 2014 Nov;146(5):673-82. doi: 10.1016/j.ajodo.2014.07.023. Epub 2014 Oct 28. PMID 25439218
- [Background] Luqmani S, Jones A, Andiappan M, Cobourne MT. A comparison of conventional vs automated digital Peer Assessment Rating scoring using the Carestream 3600 scanner and CS Model+ software system: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2020 Feb;157(2):148-155.e1. doi: 10.1016/j.ajodo.2019.10.011. PMID 32005465
- [Background] Mangano A, Beretta M, Luongo G, Mangano C, Mangano F. Conventional Vs Digital Impressions: Acceptability, Treatment Comfort and Stress Among Young Orthodontic Patients. Open Dent J. 2018 Jan 31;12:118-124. doi: 10.2174/1874210601812010118. eCollection 2018. PMID 29492177
- [Background] Mangano F, Gandolfi A, Luongo G, Logozzo S. Intraoral scanners in dentistry: a review of the current literature. BMC Oral Health. 2017 Dec 12;17(1):149. doi: 10.1186/s12903-017-0442-x. PMID 29233132
- [Background] Sivaramakrishnan G, Alsobaiei M, Sridharan K. Patient preference and operating time for digital versus conventional impressions: a network meta-analysis. Aust Dent J. 2020 Mar;65(1):58-69. doi: 10.1111/adj.12737. Epub 2019 Dec 19. PMID 31749234
- [Background] Yilmaz H, Aydin MN. Digital versus conventional impression method in children: Comfort, preference and time. Int J Paediatr Dent. 2019 Nov;29(6):728-735. doi: 10.1111/ipd.12566. Epub 2019 Aug 13. PMID 31348834